CLINICAL TRIAL: NCT05965557
Title: A Biomarker Study for Predicting the Response of Neoadjuvant Immunotherapy in Non-Small Cell Lung Cancer Based on Circulating Tumor DNA and Homologous Recombination Deficiency Analysis
Brief Title: Exploration of Predictive Markers of Neoadjuvant Immunotherapy in Non-Small Cell Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Geneplus-Beijing Co. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: PROMISEPLUS-101
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Neoadjuvant immunotherapy has become the standard perioperative treatment in lung cancer, but its effective predictive biomarkers are lacking. A small cohort reported that homologous recombination deficiency (HRD) can be used as a reliable biomarker to predict the efficacy of neoadjuvant immunotherapy, but the findings need to be validated in larger cohorts. Moreover, circulating tumor DNA (ctDNA) has the potential to predict the therapeutic efficacy of neoadjuvant immunotherapy.

This study intends to prospectively collect patients with driver-negative stage II-IIIB NSCLC who are scheduled to receive neoadjuvant immunotherapy and surgical resection and verify the value of HRD in predicting the efficacy of neoadjuvant immunotherapy. Meanwhile, the blood samples before and after neoadjuvant immunotherapy were collected for high-depth ctDNA detection to explore the correlation between the dynamic changes of ctDNA and the efficacy and prognosis of neoadjuvant immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Stage II-IIIB NSCLC
* EGFR/ALK negative
* The subjects voluntarily joined the study, signed informed consent, had good compliance, and cooperated with follow-up

Exclusion Criteria:

* A history of other malignancies within the past 5 years
* Patients with autoimmune disease are not suitable for PD1 monoclonal antibody therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage II-IIIB NSCLC who are undergoing neoadjuvant immunotherapy and surgical resection
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between HRD and MPR rate/2 years DFS | 2023/12-2025/12
  Correlation between homologous recombination deficiency (HRD) events and major pathological response (MPR) rate and DFS of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou Z, Ding Z, Yuan J, Shen S, Jian H, Tan Q, Yang Y, Chen Z, Luo Q, Cheng X, Yu Y, Niu X, Qian L, Chen X, Gu L, Liu R, Ma S, Huang J, Chen T, Li Z, Ji W, Song L, Shen L, Jiang L, Yu Z, Zhang C, Tai Z, Wang C, Chen R, Carbone DP, Xia X, Lu S. Homologous recombination deficiency (HRD) can predict the therapeutic outcomes of immuno-neoadjuvant therapy in NSCLC patients. J Hematol Oncol. 2022 May 18;15(1):62. doi: 10.1186/s13045-022-01283-7. PMID 35585646
- [Background] Provencio M, Nadal E, Insa A, Garcia-Campelo MR, Casal-Rubio J, Domine M, Majem M, Rodriguez-Abreu D, Martinez-Marti A, De Castro Carpeno J, Cobo M, Lopez Vivanco G, Del Barco E, Bernabe Caro R, Vinolas N, Barneto Aranda I, Viteri S, Pereira E, Royuela A, Casarrubios M, Salas Anton C, Parra ER, Wistuba I, Calvo V, Laza-Briviesca R, Romero A, Massuti B, Cruz-Bermudez A. Neoadjuvant chemotherapy and nivolumab in resectable non-small-cell lung cancer (NADIM): an open-label, multicentre, single-arm, phase 2 trial. Lancet Oncol. 2020 Nov;21(11):1413-1422. doi: 10.1016/S1470-2045(20)30453-8. Epub 2020 Sep 24. PMID 32979984
- [Background] Forde PM, Spicer J, Lu S, Provencio M, Mitsudomi T, Awad MM, Felip E, Broderick SR, Brahmer JR, Swanson SJ, Kerr K, Wang C, Ciuleanu TE, Saylors GB, Tanaka F, Ito H, Chen KN, Liberman M, Vokes EE, Taube JM, Dorange C, Cai J, Fiore J, Jarkowski A, Balli D, Sausen M, Pandya D, Calvet CY, Girard N; CheckMate 816 Investigators. Neoadjuvant Nivolumab plus Chemotherapy in Resectable Lung Cancer. N Engl J Med. 2022 May 26;386(21):1973-1985. doi: 10.1056/NEJMoa2202170. Epub 2022 Apr 11. PMID 35403841